CLINICAL TRIAL: NCT04038489
Title: COX Inhibition and Biomarkers of Response During Neoadjuvant Chemoendocrine Therapy for Estrogen Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Stage I-III Breast Cancer
Brief Title: COX Inhibition and Biomarkers During Neoadjuvant Chemoendocrine Therapy for ER+, HER2- Stage I-III Breast Cancer
Acronym: Breast 51
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Patrick Dillon, MD, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21822
Record Dates: First submitted 2019-07-10; First posted 2019-07-30 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer; Estrogen Receptor-positive Breast Cancer
Keywords: ER+/HER2- Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aspirin; Tamoxifen; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Intervention Model Description: All participants will receive aspirin and tamoxifen with standard AC-T chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tamoxifen and Aspirin with AC-T Chemotherapy (Experimental): AC-T chemotherapy includes 4 cycles of doxorubicin and cyclophosphamide given every 2 or 3 weeks followed by either 12 weekly cycles of lower dose paclitaxel or 4 cycles of higher dose paclitaxel every 2 or 3 weeks. During this time, all participants would receive daily aspirin and daily tamoxifen. After the AC-T chemotherapy, participants will undergo standard of care surgery to remove any remaining tumor.
  Interventions: Drug: Aspirin; Drug: Tamoxifen Pill; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Aspirin — 325 mg aspirin daily during AC-T chemotherapy
Drug: Tamoxifen Pill — Tamoxifen (either 20 mg daily or 10 mg twice a day) during AC-T chemotherapy
Drug: Doxorubicin — Doxorubicin (60 mg/m2) Given by IV with cyclophosphamide
  Other Names: Adriamycin
Drug: Cyclophosphamide — Cyclophosphamide (600 mg/m2) Given by IV with doxorubicin
  Other Names: Cytoxan
Drug: Paclitaxel — Paclitaxel 80 mg/m2 or 175 mg/m2 based on provider preference. Given by IV after completion of doxorubicin/cyclophosphamide therapy
  Other Names: Taxol

SUMMARY:
This study is designed to assess the safety and clinical activity of tamoxifen and the COX inhibitor, aspirin, given in combination with standard AC-T chemotherapy (doxorubicin, cyclophosphamide, and paclitaxel) for the treatment of high-risk estrogen receptor (ER)+, human epidermal growth factor receptor 2 (HER2)- breast cancer. If successful, the study could improve long-term outcomes for a subpopulation of women with aggressive stage I-III ER+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or older
4. Newly diagnosed with ER+/HER2- stage I-III breast cancer according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines and the 8th edition of the American Joint Committee on Cancer (AJCC); ER positive is defined as ≥ 1% positive nuclear staining
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
6. Life expectancy ≥ 6 months
7. Women of childbearing potential and men must agree to use adequate contraception (see section 5.4) prior to study entry and for at least 3 months following the last dose of tamoxifen
8. If genomic profiling has been performed (OncotypeDx, Mammaprint or other), then the score must be in a medium- or high-risk range.
9. Adequate Organ Function as described below. There are no requirements regarding recent transfusions Absolute Neutrophil Count ≥1000/mm3 Platelets ≥100,000/mm3 Hemoglobin ≥9 g/dL Serum Creatinine or Glomerular Filtration Rate (GFR) ≤ 1.5 x upper limit of normal (ULN) Bilirubin ≤ 1.5 x ULN (except in patients with Gilbert's disease, where bilirubin to 4x ULN or direct bilirubin ≤ ULN is allowed) Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN Alkaline phosphatase ≤ 2.5 x ULN
10. Ability to take oral medication

Exclusion Criteria:

1. Receipt of any systemic treatment for the current diagnosis of breast cancer (breast biopsy, excisional biopsy, or other local therapy is acceptable as long as residual disease is present and is appropriate for systemic chemotherapy and additional curative intent resection)
2. Current use of anticoagulant (e.g. warfarin (Coumadin), heparin, direct oral anticoagulants (DOAC)) within 72 hours of registration
3. Pregnancy or lactation
4. Currently in prison
5. Requirement for supplemental oxygen therapy
6. Current active cancer other than breast cancer
7. History of severe bleeding that, in the treating investigator's opinion, would put the patient at increased risk with daily 325 mg aspirin use
8. Known allergic reactions to aspirin, tamoxifen, doxorubicin, cyclophosphamide, or paclitaxel
9. Participants classified according to the New York Heart Association classification as having Class II - IV heart disease (section 12.2)
10. History of thrombosis or cerebrovascular accident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | At the time of surgery, following completion of AC-T chemotherapy, usually about 7.5 months
  Rate of participants that no longer have any tumor identified at the time of surgery after chemotherapy
Adverse events (AEs) | From time of informed consent through 30 days after completion of study intervention (for AEs) or 90 days after completion of study intervention (for Serious AEs)
  Frequency of adverse events occurring during and shortly after the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dillon, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No